CLINICAL TRIAL: NCT02794233
Title: Identification of Clinically Relevant Markers of Deep Brain Stimulation Electrode Impedance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB201600567
Record Dates: First submitted 2016-05-27; First posted 2016-06-09 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation; Electric Impedance; Parkinson disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PD patients with implanted DBS (Experimental): Impedance measurements at different time points.
  Interventions: Other: Impedance measurements

INTERVENTIONS:
Other: Impedance measurements — Refer to study description

SUMMARY:
The study will look into the changes of Deep Brain Stimulation (DBS) measured impedances in patients of Parkinson disease (PD) as a function of their functional state (lying, sitting and walking) and dopaminergic medication intake (levodopa or dopamine agonists).

The goal is to use DBS measured impedance as a surrogate of the functional and medication states of PD patients.

DETAILED DESCRIPTION:
Subjects will be recruited from the population of patients who are already implanted with DBS for treatment of PD.

At the patient's follow up visit they will be asked to come to the clinic in the "off medication" state. Off medication is defined as at least 8 hours since the last medication dosing. Data will be collected during three phases: "OFF" state, transitioning state, and "ON" state. Subjects will be asked to assume different functional states (lying, sitting or walking) for 1 minute each. During these functional states, multiple measures of impedance will be collected.

* "OFF" state data collection: The subject will be examined to assess his motor examination score using the UPDRS-III. Measurements of impedance will be collected multiple times in the lying down and sitting up states.
* Transition state data collection: The subject will be asked to take their dopamine medication. The medication will take approximately 1 hour to take full effect. Measurements of impedance will be collected every 10 minutes during this transition from the "OFF" state to the "ON" state. Patients will be asked to report at what point they felt the "ON: state (they can report the state as "OFF", "unsure", "transition" or "ON").
* "ON" state data collection: The "ON" state examination will start after 1 hour from medication administration. Subjects will be examined using the UPDRS-III. Measurements of impedance will be collected in the lying down, sitting and walking states.

Summary of the study protocol:

"OFF" state Transition state "ON' state UPDRS-III x x Impedance Lying down x x Sitting up x x x Walking x UPDRS I and II x Hoehn and Yahr x x

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's patients with DBS (unilateral or bilateral)
* Must be taking dopamine agonist or levodopa regimen
* Medtronic Neurostimulator Activa SC, PC or PC+S (IPG)

Exclusion Criteria:

* Hoehn and Yahr (H&Y) 4 and above
* History of DBS revision or lead replacement surgery
* Current or prior non-Medtronic Activa SC, PC or PC+S IPG
* Historical information of more than 1 hour delay to "ON" state as average

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-07; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in impedance value as it relates to the functional state. | 1 hour (for both outcomes)
  Functional state is defined as either: lying, sitting or walking.
Change in impedance value as it relates to the dopaminergic medication state. | 1 hour (for both outcomes)
  Dopaminergic medications are defined as either levodopa containing or dopamine agonist containing medications. The state is defined as the "OFF" state (medication effect is not present) and "ON" state (medication effect noted).

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Brito de Almeida, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Center for Movement Disorders and Neurorestoration, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Aquino CC, Fox SH. Clinical spectrum of levodopa-induced complications. Mov Disord. 2015 Jan;30(1):80-9. doi: 10.1002/mds.26125. Epub 2014 Dec 8. PMID 25488260
- [Background] Butson CR, Maks CB, McIntyre CC. Sources and effects of electrode impedance during deep brain stimulation. Clin Neurophysiol. 2006 Feb;117(2):447-54. doi: 10.1016/j.clinph.2005.10.007. Epub 2005 Dec 22. PMID 16376143
- [Background] Connolly BS, Lang AE. Pharmacological treatment of Parkinson disease: a review. JAMA. 2014 Apr 23-30;311(16):1670-83. doi: 10.1001/jama.2014.3654. PMID 24756517
- [Background] Fernandez HH. 2015 Update on Parkinson disease. Cleve Clin J Med. 2015 Sep;82(9):563-8. doi: 10.3949/ccjm.82gr.15004. PMID 26366951
- [Background] Kruk ZL, Cheeta S, Milla J, Muscat R, Williams JE, Willner P. Real time measurement of stimulated dopamine release in the conscious rat using fast cyclic voltammetry: dopamine release is not observed during intracranial self stimulation. J Neurosci Methods. 1998 Jan 31;79(1):9-19. doi: 10.1016/s0165-0270(97)00156-8. PMID 9531455
- [Background] Pandey S, Sarma N. Deep brain stimulation: current status. Neurol India. 2015 Jan-Feb;63(1):9-18. doi: 10.4103/0028-3886.152623. PMID 25751463
- [Background] Picillo M, Lozano AM, Kou N, Munhoz RP, Fasano A. Programming Deep Brain Stimulation for Tremor and Dystonia: The Toronto Western Hospital Algorithms. Brain Stimul. 2016 May-Jun;9(3):438-452. doi: 10.1016/j.brs.2016.02.003. Epub 2016 Feb 12. PMID 26968805
- [Background] Satzer D, Maurer EW, Lanctin D, Guan W, Abosch A. Anatomic correlates of deep brain stimulation electrode impedance. J Neurol Neurosurg Psychiatry. 2015 Apr;86(4):398-403. doi: 10.1136/jnnp-2013-307284. Epub 2014 Jun 16. PMID 24935985